CLINICAL TRIAL: NCT06238557
Title: Prospective Evaluation of Psychological Consequences and Impact on Long-term Quality of Life
Acronym: PICS
Status: Completed | Type: Observational
Sponsor: Romain Ronfle (Other)
Responsible Party: Sponsor-Investigator, Romain Ronfle, Principal investigator, Centre Hospitalier Intercommunal Aix-Pertuis
Organization: Centre Hospitalier Intercommunal Aix-Pertuis (Other)
Other Study IDs: 20220205-7
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Quality of Life; Post ICU Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to show the patient discomfort during their stay in intensive care is directly linked to the occurrence of a post ICU syndrome at 3 months.

The main questions it aims to answer are :

* Evaluate the value of the IPREA score on quality of life impairment a 3 months ;
* Identify the 3 areas of discomfort most associated with progression to a post ICU syndrome at 3 months ;
* Define a threshold value for the IPREA score ;
* Correlate clinical assessment and psychological follow-up with the to the prediction of a post ICU syndrome ;
* Establish a correlation between IPREA score and time to first rise
* Establish a correlation between identified factors of post ICU syndrome and IPREA score

DETAILED DESCRIPTION:
A stay in intensive care can be seen as a stressful ordeal for a patient's body, both physically and morally. Among patients alive following a stay in intensive care, half have a disabling psychiatric disorder. The main psychiatric disorders described in post-resuscitation are anxiety, depression and post-traumatic stress disorder (PTSD). When one of these disorders is present, there is a 64% chance that it will coexist with one of the other two disorders. These psychological disorders will have an impact on the quality of life and mortality of patients leaving intensive care. Depression is independently associated with an increased risk of further hospitalisation. These different psychological and somatic disorders can be found in the same entity: post-resuscitation syndrome (PRS).

In a context where the proportion of awake patients is growing in our intensive care units, the impact of subjective factors is becoming increasingly important. A stay in intensive care is marked by a stressful environment for the patient at several levels, as well as by care procedures that are often experienced as traumatic (mechanical ventilation, dialysis and invasive procedures). For example, memories of terrifying experiences, often the source of nightmares or hallucinations that persist beyond the hospital stay, encourage the development of PTSD. Similarly, certain environmental factors such as lighting conditions and noise levels can have an impact on patient comfort during their stay in intensive care, confirming the importance of better controlling all external factors that can contribute to stress. Targeted measures centred on an isolated objective, such as reducing thirst, have shown real clinical benefit in terms of patient outcome. Recognition of these sources of discomfort in intensive care and resuscitation units is a first step towards optimising patient comfort. A research team have developed a standardised and validated discomfort score (Discomforts of Patients in Intensive Care, IPREA) that enables several discomforts perceived throughout the intensive care stay to be identified and quantified.

In addition to the psychiatric consequences, the investigators know that patients who survive a stay in intensive care face physical and cognitive consequences for their state of health. PRS is a concept that includes these three dimensions, defined as cognitive dysfunction, acquired physical weakness and altered mental health. It is thought to affect at least 50% of patients. The growing interest in this syndrome is explained by its multi-dimensional aspect, which is representative of patients' long-term quality of life. The potential impact between discomfort in intensive care and long-term psychiatric consequences, or more broadly the occurrence of an PRS, is a central question with an impact on our daily practice. In addition, a bedside assessment using simple tools as part of a psychological follow-up could help to prevent or at least recognise early the factors favouring an PRS.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the intensive care unit at Aix-en-Provence hospital (sepsis, acute respiratory distress, disturbed consciousness, emergency surgery, etc.)
* Minimum stay of 3 calendar days

Exclusion Criteria:

* Patient under 18 years
* Patients deprived of their liberty, under guardianship or trusteeship
* Non-French-speaking patient
* Presence of a pre-existing cognitive disorder as assessed by a clinician
* Participation in an interventional research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU during minimum 3 days
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-10-14 (Actual)

PRIMARY OUTCOMES:
Assessing the impact of the overall discomfort of intensive care patients on the occurrence of a psychiatric RPD at 3 months | 3 months
  Occurrence of discomfort in intensive care as defined by the IPREA score

SECONDARY OUTCOMES:
Assessing the value of the IPREA score in terms of quality of life at 3 months | 3 months
  Relation between IPREA score and quality of life
Identifying the 3 areas of discomfort most associated with progression to post ICU syndrome at 3 months | 3 months
  Relation between discomfort during hospitalization and post ICU syndrome
Defining a threshold value for the IPREA score | through study completion, an average of 1 year
  Evaluation of IPREA score
Correlation between clinical assessment and psychological follow-up with the post ICU syndrome | through study completion, an average of 1 year
  Clinical experience of the clinician and the psychologist and the interest in predicting a post ICU syndrome
Establish a correlation between IPREA score and time to first rise | through study completion, an average of 1 year
  Evaluation of IPREA score
Correlation between identified factors of post ICU syndrome and IPREA score | through study completion, an average of 1 year
  Evaluation and relation between factors of post ICU syndrome and IPREA score

CONTACTS AND LOCATIONS:
Overall Officials: Romain RONFLE, MD, Principal Investigator — Centre Hospitalier Intercommunal Aix-Pertuis
Locations (1):
- Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence, France